CLINICAL TRIAL: NCT04012034
Title: Treatment With Punction and Radiofrequency of Active Trigger Points in Patients With Pelvic Chronic Pain and History of Endometriosis
Brief Title: Treatment With Radiofrequency in Patients With Chronic Pelvic Pain and History of Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Francisco Carmona, Head of gynecology department, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RFDP
Record Dates: First submitted 2019-05-25; First posted 2019-07-09 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Endometriosis; Chronic Pain; Quality of Life
MeSH Terms: conditions — Endometriosis; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency A (Experimental): Treatment with radiofrequency
  Interventions: Device: Radiofrequency A
- Placebo (Placebo Comparator): Treatment with radiofrequency without energy
  Interventions: Device: Radiofrequency B

INTERVENTIONS:
Device: Radiofrequency A — Application of radiofrequency for 30 minutes per week during 8 weeks
  Arms: Radiofrequency A
Device: Radiofrequency B — Application of radiofrequency without energy for 30 minutes per week during 8 weeks
  Arms: Placebo

SUMMARY:
Managing chronic pelvic pain in patients with a past history of endometriosis might be a challenge for the gynaecologist.

The objective of this study is to evaluate pelvic pain after treatment with radiofrequency in patients with chronic pelvic pain and surgery for endometriosis.

DETAILED DESCRIPTION:
Patients with pelvic chronic pain and a past history of endometriosis without imaging evidence of endometriosis in the present will be enrolled in this study. The main objective of this study is to evaluate improvement of pelvic pain these patients. Moreover, quality of life and sexual function will be also assessed. Patients who are enrolled will come once a week per eight weeks to the hospital to have 30 minutes treatment with radiofrequency. They will be randomised in two groups, one receiving the radiofrequency and the other not (the device will be not give the energy). At the enrollement visit, the SF-36, VAS score, anxiety and depression tests and sexual function tests will be answered the patients. At the end of the treatment, and one month after the end, they will answer the same questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pelvic pain
* Past surgery for endometriosis

Exclusion Criteria:

* Active endometriosis, diagnosed by imaging techniques
* Presence of other diseases that can cause chronic pelvic pain
* Contraindication for the radiofrequency use: pregnancy, metallic prothesis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain: VAS score | Baseline (Before starting the study)
  Visual Analogue Scale Score, from 0 to 10, where 0 is no pain at all and 10 is the worst pain ever.
Pain: VAS score | 1 month after study completion
  Visual Analogue Scale Score, from 0 to 10, where 0 is no pain at all and 10 is the worst pain ever.

SECONDARY OUTCOMES:
Quality of life: QoL SF-36 | Before starting the study
  QoL SF-36, scale where 0 is maximum disability and a score of 100 is equivalent to no disability
Quality of life: QoL SF-36 | 1 month after study completion
  QoL SF-36, scale where 0 is maximum disability and a score of 100 is equivalent to no disability
Female Sexual Function Index (FSFI) | Before starting the study
  Female Sexual Function Index (FSFI), minimum score is 2 and maximum score is 36, meaning no disfunction at all
Female Sexual Function Index (FSFI) | 1 month after study completion
  Female Sexual Function Index (FSFI), minimum score is 2 and maximum score is 36, meaning no disfunction at all

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Carmona, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
It is not intended to share IPD to other researchers since it is the first study of this kind in our setting.